CLINICAL TRIAL: NCT01361763
Title: Phase II, Randomized, Crossover, Single Blind, Safety Trial of DABIGATRAN Versus ASA for Preventing Ischaemic Brain Lesions in Patients Affected by CADASIL
Brief Title: Safety Study of Dabigatran in CADASIL
Acronym: SONICA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Francesco Orzi, Department of Neuroscience, Mental Healt and Sensory Organs (NESMOS); University of Rome "La Sapienza"
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DABCAD2010
Record Dates: First submitted 2011-05-16; First posted 2011-05-27 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: CADASIL
Keywords: Dabigatran; Microbleeds; Microthrombi; CADASIL; Small Vessel Disease
MeSH Terms: conditions — CADASIL | interventions — Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dabigatran (Experimental)
  Interventions: Drug: Dabigatran
- Antiplatelets (Active Comparator)
  Interventions: Drug: Antiplatelets

INTERVENTIONS:
Drug: Dabigatran — 110 mg twice daily
  Arms: Dabigatran
Drug: Antiplatelets — 100mg once a day
  Arms: Antiplatelets

SUMMARY:
This study is a Phase II, randomized, crossover trial designed to compare one fixed dose of dabigatran with open-label use of ASA in patients affected by CADASIL; the study is a safety trial, and the primary objective is to assess that dabigatran is not less safe than ASA in subjects with CADASIL.

DETAILED DESCRIPTION:
The primary endpoint is the number of microbleeds, as measured by MRI, at 90 days of follow up.

The study is based on the hypothesis that drugs inhibitor of the thrombin is more effective than ASA in preventing vessel obstruction. The rationale behind the study is based on the assumption that: a) the formation of microthrombi is relevant to the clinical expression of the CADASIL disease, and b) thrombin inhibitors are more effective than antiplatelet drugs in preventing lesions by microvessel obstruction.

Eligible patients will be randomized into one of the 2 treatment groups:

1. One week wash-out (W1), Dabigatran one tablet 100mg twice a day for 12 weeks, a second one week wash-out (W2), treatment with ASA one tablet of 100mg/day once a day for 12 weeks;
2. The same scheme repeated with reversed sequence No initial wash-out week will be required for patients in group 2 already treated with ASA.

Clinical and instrumental evaluations will be carried out during the first (W1) and second wash-out weeks (W2), and at the end of the study (during the week that follows the second treatment regimen (W3). Each evaluation will consist of physical examination, blood tests and MRI.

Safety is evaluated on the basis of brain microbleeds and severe haemorrhages.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed with CADASIL according genetic test will be eligible.

Exclusion Criteria:

* Treatment with antiplatelet drugs for a condition different from CADASIL;
* conditions associated with an increased risk of bleeding (major surgery within the previous month, planned surgery or intervention within the next 3 months;
* history of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding;
* gastrointestinal hemorrhage within the past year;
* symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days; hemorrhagic disorder or bleeding diathesis;
* need for anticoagulant treatment of disorders other than atrial fibrillation; fibrinolytic agents within 48 hours of study entry; uncontrolled hypertension (systolic blood pressure greater than 180 mm Hg and/or diastolic blood pressure greater than 100 mm Hg);
* recent malignancy or radiation therapy (within 6 months) and not expected to survive 3 years; severe renal impairment (estimated creatinine clearance 30 mL/min or less);
* active infective endocarditis;
* active liver disease (including but not limited to persistent ALT, AST, Alk Phos greater than twice the upper limit of the normal range; active hepatitis C (positive HCV RNA);
* active hepatitis B (HBs antigen +, anti HBc IgM +), active hepatitis A);
* women who are pregnant or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Number of microbleeds on MRI | Six Months
  Primary endpoint is defined as the difference in number of microbleeds on MRI images taken at the end of the 2 treatments (i.e, during W2 and W3). Secondary endpoint is major bleeding. The neuroradiologists (or trained neurologists) who will examine the images on MRI will be blind to treatment.

SECONDARY OUTCOMES:
Major bleeding | Six Months
  Severe haemorrhages are defined as a reduction of the haemoglobin level by at least 20g per litre, need of a transfusion of at least 2 units of blood, or symptomatic bleeding of an organ or critical area. Life threatening haemorrhages are a subcategory of severe hemorrhages defined as: fatal haemorrhages, symptomatic intracranial haemorrhages, haemorrhages with a diminution of haemoglobin level of at least 50g per litre or that require transfusion of at least 4 blood units, or surgery. All the other haemorrhages are considered minor.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orzi, MD, Study Chair — NESMOS Department, University of Rome "La Sapienza"; St. Andrea Hospital
Locations (2):
- Italy (2):
  - Emergency Department Stroke Unit, Umberto I Hospital, Rome, Rome
  - NESMOS Department St. Andrea Hospital, Rome, Rome

REFERENCES:
- [Background] Bailey EL, McCulloch J, Sudlow C, Wardlaw JM. Potential animal models of lacunar stroke: a systematic review. Stroke. 2009 Jun;40(6):e451-8. doi: 10.1161/STROKEAHA.108.528430. Epub 2009 Apr 23. PMID 19390080
- [Background] Chen B, Cheng Q, Yang K, Lyden PD. Thrombin mediates severe neurovascular injury during ischemia. Stroke. 2010 Oct;41(10):2348-52. doi: 10.1161/STROKEAHA.110.584920. Epub 2010 Aug 12. PMID 20705928
- [Background] Chabriat H, Joutel A, Dichgans M, Tournier-Lasserve E, Bousser MG. Cadasil. Lancet Neurol. 2009 Jul;8(7):643-53. doi: 10.1016/S1474-4422(09)70127-9. PMID 19539236
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Cumurciuc R, Guichard JP, Reizine D, Gray F, Bousser MG, Chabriat H. Dilation of Virchow-Robin spaces in CADASIL. Eur J Neurol. 2006 Feb;13(2):187-90. doi: 10.1111/j.1468-1331.2006.01113.x. PMID 16490051
- [Background] Dichgans M, Holtmannspotter M, Herzog J, Peters N, Bergmann M, Yousry TA. Cerebral microbleeds in CADASIL: a gradient-echo magnetic resonance imaging and autopsy study. Stroke. 2002 Jan;33(1):67-71. doi: 10.1161/hs0102.100885. PMID 11779891
- [Background] Heye N, Paetzold C, Steinberg R, Cervos-Navarro J. The topography of microthrombi in ischemic brain infarct. Acta Neurol Scand. 1992 Nov;86(5):450-4. doi: 10.1111/j.1600-0404.1992.tb05122.x. PMID 1481626
- [Background] Hills M, Armitage P. The two-period cross-over clinical trial. Br J Clin Pharmacol. 1979 Jul;8(1):7-20. doi: 10.1111/j.1365-2125.1979.tb05903.x. No abstract available. PMID 552299
- [Background] Bokura H, Kobayashi S, Yamaguchi S. Distinguishing silent lacunar infarction from enlarged Virchow-Robin spaces: a magnetic resonance imaging and pathological study. J Neurol. 1998 Feb;245(2):116-22. doi: 10.1007/s004150050189. PMID 9507419
- [Background] Oh JH, Lee JS, Kang SY, Kang JH, Choi JC. Aspirin-associated intracerebral hemorrhage in a patient with CADASIL. Clin Neurol Neurosurg. 2008 Apr;110(4):384-6. doi: 10.1016/j.clineuro.2007.12.001. Epub 2008 Jan 22. PMID 18207319
- [Background] Kario K, Matsuo T, Hoshide S, Umeda Y, Shimada K. Effect of thrombin inhibition in vascular dementia and silent cerebrovascular disease. An MR spectroscopy study. Stroke. 1999 May;30(5):1033-7. doi: 10.1161/01.str.30.5.1033. PMID 10229740
- [Background] Lesnik Oberstein SA, van den Boom R, van Buchem MA, van Houwelingen HC, Bakker E, Vollebregt E, Ferrari MD, Breuning MH, Haan J; Dutch CADASIL Research Group. Cerebral microbleeds in CADASIL. Neurology. 2001 Sep 25;57(6):1066-70. doi: 10.1212/wnl.57.6.1066. PMID 11571335
- [Background] Pfefferkorn T, von Stuckrad-Barre S, Herzog J, Gasser T, Hamann GF, Dichgans M. Reduced cerebrovascular CO(2) reactivity in CADASIL: A transcranial Doppler sonography study. Stroke. 2001 Jan;32(1):17-21. doi: 10.1161/01.str.32.1.17. PMID 11136908
- [Background] Rouhl RP, van Oostenbrugge RJ, Knottnerus IL, Staals JE, Lodder J. Virchow-Robin spaces relate to cerebral small vessel disease severity. J Neurol. 2008 May;255(5):692-6. doi: 10.1007/s00415-008-0777-y. Epub 2008 Feb 21. PMID 18286319
- [Background] Stenborg A, Kalimo H, Viitanen M, Terent A, Lind L. Impaired endothelial function of forearm resistance arteries in CADASIL patients. Stroke. 2007 Oct;38(10):2692-7. doi: 10.1161/STROKEAHA.107.490029. Epub 2007 Aug 30. PMID 17761910
- [Background] Turturro F, Rocca B, Gumina S, De Cristofaro R, Mangiola F, Maggiano N, Evangelista A, Salsano V, Montanaro A. Impaired primary hemostasis with normal platelet function in Duchenne muscular dystrophy during highly-invasive spinal surgery. Neuromuscul Disord. 2005 Aug;15(8):532-40. doi: 10.1016/j.nmd.2005.05.005. PMID 16009551
- [Background] van Den Boom R, Lesnik Oberstein SA, van Duinen SG, Bornebroek M, Ferrari MD, Haan J, van Buchem MA. Subcortical lacunar lesions: an MR imaging finding in patients with cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy. Radiology. 2002 Sep;224(3):791-6. doi: 10.1148/radiol.2243011123. PMID 12202716
- [Background] Wang CX, Ding X, Shuaib A. Treatment with melagatran alone or in combination with thrombolytic therapy reduced ischemic brain injury. Exp Neurol. 2008 Sep;213(1):171-5. doi: 10.1016/j.expneurol.2008.05.020. Epub 2008 Jun 7. PMID 18598697
- [Background] Yin X, Wright J, Wall T, Grammas P. Brain endothelial cells synthesize neurotoxic thrombin in Alzheimer's disease. Am J Pathol. 2010 Apr;176(4):1600-6. doi: 10.2353/ajpath.2010.090406. Epub 2010 Feb 11. PMID 20150433
- [Background] Mastroiacovo F, Busceti CL, Biagioni F, Moyanova SG, Meisler MH, Battaglia G, Caricasole A, Bruno V, Nicoletti F. Induction of the Wnt antagonist, Dickkopf-1, contributes to the development of neuronal death in models of brain focal ischemia. J Cereb Blood Flow Metab. 2009 Feb;29(2):264-76. doi: 10.1038/jcbfm.2008.111. Epub 2008 Oct 1. PMID 18827832
- [Background] Zhang QG, Wang R, Khan M, Mahesh V, Brann DW. Role of Dickkopf-1, an antagonist of the Wnt/beta-catenin signaling pathway, in estrogen-induced neuroprotection and attenuation of tau phosphorylation. J Neurosci. 2008 Aug 20;28(34):8430-41. doi: 10.1523/JNEUROSCI.2752-08.2008. PMID 18716201
- [Background] Rosi MC, Luccarini I, Grossi C, Fiorentini A, Spillantini MG, Prisco A, Scali C, Gianfriddo M, Caricasole A, Terstappen GC, Casamenti F. Increased Dickkopf-1 expression in transgenic mouse models of neurodegenerative disease. J Neurochem. 2010 Mar;112(6):1539-51. doi: 10.1111/j.1471-4159.2009.06566.x. Epub 2009 Dec 29. PMID 20050968
- [Background] De Ferrari GV, Moon RT. The ups and downs of Wnt signaling in prevalent neurological disorders. Oncogene. 2006 Dec 4;25(57):7545-53. doi: 10.1038/sj.onc.1210064. PMID 17143299